CLINICAL TRIAL: NCT00990223
Title: A Phase 1, Double-Blind (Sponsor Open), Randomized, Placebo-Controlled Trial To Evaluate The Effects Of 100 MG Once Daily Of Eplerenone On Serum Aldesterone And Plasma Renin Activity During 10 Days Of Dosing In Healthy Volunteers
Brief Title: Effects Of Eplerenone On Serum Aldesterone And Plasma Renin Activity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Other
Other Study IDs: A6141115
Record Dates: First submitted 2009-10-05; First posted 2009-10-06 (Estimated); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Healthy Volunteers
Keywords: Eplerenone Aldosterone and Plasma Renin Activity responses Pharmacodynamics
MeSH Terms: interventions — Eplerenone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cohort 1 (Experimental): Healthy Volunteers - eplerenone versus placebo.
  Interventions: Drug: Eplerenone or Placebo

INTERVENTIONS:
Drug: Eplerenone or Placebo — Eplerenone 100 mg or Placebo, daily for 10 days.

SUMMARY:
To evaluate the changes in serum aldosterone and plasma renin activity on Day 0 and on Days 1 and 10 after administration of 100 mg of eplerenone daily for 10 days.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs)
* Subjects who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

* Evidence or history of clinically significant disease
* Subjects with a supine BP greater than or equal to 140 mm Hg systolic or greater than or equal to 90 mm Hg diastolic or <100 mm Hg systolic and <60 mm Hg diastolic on a single measurement, as described in the protocol
* Blood donation of approximately 1 pint (500 mL) within 56 days prior to dosing
* History of sensitivity to eplerenone, spironolactone or related compounds.
* Serum potassium >5.0 mEq/L at screening or Day 0

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2009-10; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Area under the effect curve (AUEC) for serum aldosterone and PRA on Day 0 and on Days 1 and 10 after administration of 100 mg of eplerenone | 11 days

SECONDARY OUTCOMES:
Single Dose PK for eplerenone: Cmax, Tmax, and AUCtau; Multiple Dose PK for eplerenone: Cmax(ss), Tmax(ss), AUC(,tau,ss), half life, Cmin(ss), Cave(ss), accumulation ratios AUC(tau,ss)/AUC(tau,sd) and Cmax(ss)/Cmax(sd). | 13 days
Safety and tolerability of eplerenone as determined by adverse event reporting, clinical laboratory results, vital signs (supine blood pressure and heart rate), physical examinations and ECGs. | 13 days
Change from baseline (Day 0) to Day 8 in exploratory mRNA gene expression biomarkers (SGK1: Serum/glucocorticoid regulated kinase 1 gene, ENaCα: Epithelial Sodium Channel alpha subunit, ENaCγ: Epithelial Sodium Channel gamma subunit, | 9 days
MR: Mineralcorticoid Receptor, ACTβ: Beta Actin) after administration of eplerenone or placebo. These results will not be included in the study report. | 9 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- United States (2):
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, South Miami, Florida

REFERENCES:
- [Derived] Eudy RJ, Sahasrabudhe V, Sweeney K, Tugnait M, King-Ahmad A, Near K, Loria P, Banker ME, Piotrowski DW, Boustany-Kari CM. The use of plasma aldosterone and urinary sodium to potassium ratio as translatable quantitative biomarkers of mineralocorticoid receptor antagonism. J Transl Med. 2011 Oct 21;9:180. doi: 10.1186/1479-5876-9-180. PMID 22017794
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6141115&StudyName=Effects%20Of%20Eplerenone%20On%20Serum%20Aldesterone%20And%20Plasma%20Renin%20Activity